CLINICAL TRIAL: NCT03547245
Title: A Phase 1, Randomized, Double-blind, Placebo-controlled Dosage Escalation Trial to Evaluate the Safety and Immunogenicity of eOD-GT8 60mer Vaccine, Adjuvanted in HIV-uninfected, Healthy Adult Volunteers
Brief Title: A Phase I Trial to Evaluate the Safety and Immunogenicity of eOD-GT8 60mer Vaccine, Adjuvanted
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: International AIDS Vaccine Initiative (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: G001
Record Dates: First submitted 2018-04-27; First posted 2018-06-06 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HIV-uninfected, healthy adults (Active Comparator)
  Interventions: Biological: eOD-GT8 60mer + AS01B/ DPBS sucrose/IM; Biological: DPBS Sucrose
- HIV-uninfected, healthy adults - placebo (Placebo Comparator)
  Interventions: Biological: DPBS Sucrose

INTERVENTIONS:
Biological: eOD-GT8 60mer + AS01B/ DPBS sucrose/IM — 20 μg
  Arms: HIV-uninfected, healthy adults
Biological: eOD-GT8 60mer + AS01B/ DPBS sucrose/IM — 100 μg
  Arms: HIV-uninfected, healthy adults
Biological: DPBS Sucrose — Placebo

SUMMARY:
This is a phase 1 first-in-human clinical trial to assess the safety, tolerability, and immunogenicity of eOD-GT8 60mer Vaccine, Adjuvanted, in up to 48 healthy adult HIV-negative volunteers.

DETAILED DESCRIPTION:
This is a phase 1 first-in-human clinical trial to assess the safety, tolerability, and immunogenicity of eOD-GT8 60mer Vaccine, Adjuvanted, in up to 48 healthy adult HIV-negative volunteers. The study is a randomized, double-blind, placebo-controlled dosage-escalation Phase 1 study intended to evaluate the safety and immunogenicity of eOD-GT8 60mer Vaccine, Adjuvanted in a prime-boost regimen.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female, including transgender individuals, as assessed by a medical history, physical exam, and laboratory tests;
2. At least 18 years of age on the day of screening and has not reached his/her 51st birthday on the day of first IP administration;
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study;
4. In the opinion of the Principal Investigator or designee and based on Assessment of Informed Consent Understanding results, has understood the information provided and potential impact and/or risks linked to vaccination and participation in the trial; written informed consent will be obtained from the volunteer before any study-related procedures are performed;
5. Willing to undergo HIV testing, risk reduction counseling and receive HIV test result;
6. All heterosexually active female volunteers must commit to use an effective method of contraception for 4 months following investigational product administration
7. All female volunteers must be willing to undergo urine pregnancy tests at time points indicated in the Schedule of Procedures and must test negative prior to each study vaccination;
8. All sexually active males (unless anatomically sterile or in a monogamous relationship with a female partner who uses a documented non-barrier method of birth control) must be willing to use an effective method of contraception (such as consistent condom use) from the day of first vaccination until at least 4 months after the last vaccination ;
9. Willing to forgo donations of blood, or any other tissues during the study and, for those who test HIV-positive due to vaccine-induced antibodies, until the anti-HIV antibody titers become undetectable;
10. Women, who are not heterosexually active at screening, must agree to utilize an effective method of contraception if they become hetero-sexually active, as outlined above.

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection; any clinically relevant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids (the use of topical, nasal or inhaled steroids is permitted), immunosuppressive, anticancer, anti-tuberculosis or other medications considered significant by the investigator within the previous 6 months;
2. The following exceptions are permitted and will not exclude study participation: use of corticosteroid nasal spray for rhinitis, topical corticosteroids for an acute uncomplicated dermatitis; or a short course (duration of 10 days or less, or a single injection) of corticosteroid for a non-chronic condition (based on investigator clinical judgment) at least 2 weeks prior to enrollment in this study;
3. Any clinically significant acute or chronic medical condition that is considered progressive or in the opinion of the investigator makes the volunteer unsuitable for participation in the study;
4. Reported risky behavior for HIV infection within 12 months prior to vaccination
5. If female, pregnant or planning a pregnancy during the period of enrollment until 4 months after the last study vaccination; or lactating;
6. Bleeding disorder that was diagnosed by a physician (e.g., clotting factor deficiency, coagulopathy or platelet disorder that requires special precautions) (Note: A volunteer who states that he or she has easy bruising or bleeding, but does not have a formal diagnosis and has had IM vaccine administrations and blood draws without any adverse experience, is eligible);
7. Infectious disease: chronic hepatitis B infection (HbsAg-positive), current hepatitis C infection (HCV Ab positive and HCV RNA positive) treatment for chronic hepatitis C infection in the past year, or active syphilis (positive RPR confirmed by TPHA);
8. Receipt of live attenuated vaccine within the previous 30 days or planned receipt within 30 days after vaccination with Investigational Product; or receipt of other vaccine within the previous 14 days or planned receipt within 14 days after vaccination with Investigational Product. (Exception is live attenuated influenza vaccine within 14 days);
9. History of splenectomy;
10. Receipt of blood transfusion or blood-derived products within the previous 3 months;
11. Any of the following abnormal laboratory parameters listed below:

    Hematology
    * Hematocrit: <35%
    * Absolute Neutrophil Count (ANC): ≤1,000/mm3
    * Absolute Lymphocyte Count (ALC): ≤650/mm3
    * Platelets: <125,000 cells/mm3 Chemistry
    * Creatinine >1.1 x upper limit of normal (ULN)
    * ALT >1.25 x ULN
    * AST >1.25 x ULN Urinalysis
    * Clinically significant abnormal dipstick confirmed by microscopy:
    * Protein = 1+ or more
    * Blood = 2+ or more (not due to menses)
12. Participation in another clinical trial of an Investigational Product currently, within the previous 3 months or expected participation during this study (Concurrent participation in an observational trial not requiring any blood or tissue sample collection is not an exclusion);
13. Prior receipt of another investigational HIV vaccine candidate (Note: receipt of placebo in a previous HIV vaccine trial will not exclude a volunteer from participation if documentation is available and the Medical Monitor gives approval);
14. History of severe local or systemic reactogenicity to vaccines (e.g., anaphylaxis, respiratory difficulties, angioedema, injection site necrosis or ulceration);
15. Psychiatric condition that compromises safety of the volunteer and precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years (prior to screening), ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years;
16. Seizure disorder: A volunteer who has had a seizure in the last 3 years (prior to screening) is excluded. (Not excluded: a volunteer with a history of seizures who has neither required medications nor had a seizure for 3 years);
17. A history of malignancy in the past 5 years (prior to screening) or ongoing malignancy (A history of a completely excised malignancy that is considered cured is not an exclusion);
18. Active, serious infections requiring parenteral antibiotic, antiviral or antifungal therapy within 30 days prior to enrollment;
19. Body mass index ≥35 ;
20. Body weight <110 pounds (55 kg);
21. If, in the opinion of the Principal Investigator, it is not in the best interest of the volunteer to participate in the trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2021-08-13 (Actual)

PRIMARY OUTCOMES:
Safety and Tolerability: frequency of local and systemic reactogenicity events | 7 days
  To evaluate the safety and tolerability of the study regimens based on the frequency of local and systemic reactogenicity events as assessed using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (v2.1).
Safety and Tolerability: proportion of volunteers with moderate or greater unsolicited adverse events | 16 months
  To evaluate the safety and tolerability of the study regimens based on the proportion of volunteers with moderate or greater unsolicited adverse events including safety laboratory as assessed using the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (v2.1).
Safety and Tolerability: proportion of volunteers in each group with potential immune-mediated diseases (pIMDs) | 16 months
  To evaluate the proportion of volunteers in each group with potential immune-mediated diseases (pIMDs) based on a defined list of pIMDs in the study protocol.

SECONDARY OUTCOMES:
Immunogenicity: Frequency of responses | 16 months
  To evaluate the frequency of eOD-GT8 60mer-specific, eOD-GT8 monomer-specific, and epitope-specific serum antibody responses after 1st and/or 2nd immunization compared to baseline and placebo
Immunogenicity: Magnitude of responses | 16 months
  To evaluate the magnitude of eOD-GT8 60mer-specific, eOD-GT8 monomer-specific, and epitope-specific serum antibody responses after 1st and/or 2nd immunization compared to baseline and placebo

CONTACTS AND LOCATIONS:
Overall Officials: David Diemert, MD, FRCP(C), Principal Investigator — George Washington University School of Medicine & Health Sciences; Julie McElrath, MD, PhD, Principal Investigator — Seattle HIV Vaccine Trials Unit
Locations (2):
- United States (2):
  - George Washington University, Washington D.C., District of Columbia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington

REFERENCES:
- [Derived] Yan H, Peng Y, Zhang J, Peng R, Feng X, Su J, Yi H, Lu Y, Gao S, Liu J, Yang M, Liu X, Gao S, Chen Z. Rapid and highly potent humoral responses to mpox nanovaccine candidates adjuvanted by thermostable scaffolds. Vaccine. 2024 Mar 19;42(8):2072-2080. doi: 10.1016/j.vaccine.2024.02.027. Epub 2024 Feb 28. PMID 38423815
- See also: Related Info — http://iavi.org